CLINICAL TRIAL: NCT03160898
Title: A Phase 2, Multi-Center, Double-Blind, Randomized, Dose-Ranging, Placebo-Controlled Study to Evaluate the Efficacy, Safety and Tolerability of CK-2127107 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: A Study to Evaluate Efficacy, Safety and Tolerability of CK-2127107 in Patients With Amyotrophic Lateral Sclerosis (ALS)
Acronym: FORTITUDE-ALS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CY 5022
Record Dates: First submitted 2017-05-12; First posted 2017-05-19 (Actual); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; CK-2127107; Reldesemtiv
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — reldesemtiv

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Reldesemtiv 150 mg twice daily (Experimental): Patients in this arm took 1 reldesemtiv 150 mg oral tablet and 2 matching placebo tablets every 12 hours for 12 weeks.
  Interventions: Drug: Reldesemtiv
- Reldesemtiv 300 mg twice daily (Experimental): Patients in this arm took 2 reldesemtiv 150 mg oral tablets and 1 matching placebo tablet every 12 hours for 12 weeks.
  Interventions: Drug: Reldesemtiv
- Reldesemtiv 450 mg twice daily (Experimental): Patients in this arm took 3 reldesemtiv 150 mg oral tablets every 12 hours for 12 weeks.
  Interventions: Drug: Reldesemtiv
- Placebo (Placebo Comparator): Patients in this arm took 3 placebo oral tablets every 12 hours for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Reldesemtiv — Oral tablet
  Other Names: CK-2127107
  Arms: Reldesemtiv 150 mg twice daily; Reldesemtiv 300 mg twice daily; Reldesemtiv 450 mg twice daily
Drug: Placebo — Oral tablet
  Arms: Placebo

SUMMARY:
The purpose of this study was to assess the effect of CK-2127107 (hereafter referred to as reldesemtiv) versus placebo on respiratory function and other measures of skeletal muscle function in patients with ALS.

DETAILED DESCRIPTION:
This was a double-blind, randomized, placebo-controlled, dose ranging study of reldesemtiv in patients with ALS. Eligible patients were randomized (1:1:1:1) to receive placebo or one of three doses of reldesemtiv (150, 300, or 450 mg twice daily) for 12 weeks. Randomization was stratified by riluzole concomitant use/non-use and edaravone concomitant use/non-use. Concomitant riluzole and edaravone were allowed as long as the riluzole dose had been stable for at least 30 days prior to screening and edaravone had been taken for 2 cycles prior to screening; these drugs could not be initiated during the study.

A total of 7 study visits were planned: screening, Day 1 (first dosing day), Weeks 2, 4, 8, and 12, and follow-up (4 weeks after the last dose of study drug). Study drug (placebo or reldesemtiv) was to be taken twice daily, approximately 12 hours (± 2 hours) apart and within 2 hours following a meal.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of familial or sporadic ALS ≤ 24 months prior to screening
* Upright Slow Vital Capacity (SVC) ≥ 60% of predicted for age, height and sex at screening
* Able to swallow tablets
* A caregiver (if one is needed)
* Able to perform reproducible pulmonary function tests
* Pre-study clinical laboratory findings within the normal range or, if outside the normal range, deemed not clinically significant by the Investigator
* Male patients who have not had a vasectomy and confirmed zero sperm count must agree after receiving the first dose of study drug until 10 weeks after the last dose to either use acceptable methods of contraception or abstain from sex
* Female patients must be post-menopausal or sterilized or must not be breastfeeding, have a negative pregnancy test, have no intention to become pregnant during the study and use acceptable methods of contraception or abstain from heterosexual intercourse from Screening until 10 weeks after last dose of study drug
* Patients must be either on riluzole for at least 30 days prior to screening or have not taken riluzole for at least 30 days prior to screening and not planning to start riluzole during the course of the study.
* Patients on edaravone must have completed at least 2 cycles of dosing with edaravone at the time of screening or have not taken edaravone for at least 30 days prior to screening and not planning to start edaravone during the course of the study.

Exclusion Criteria:

* At the time of screening, any use of non-invasive ventilation (NIV), e.g. continuous positive airway pressure [CPAP], noninvasive bi-level positive airway pressure [NPPV] or noninvasive volume ventilation [NVV] for any portion of the day, or mechanical ventilation via tracheostomy, or on any form of oxygen supplementation
* Neurological impairment due to a condition other than ALS
* Presence at screening of any medically significant cardiac, pulmonary, GI, musculoskeletal, or psychiatric illness that might interfere with the patient's ability to comply with study procedures or that might confound the interpretation of clinical safety or efficacy data
* Has taken any investigational study drug within 30 days or five half-lives of the prior agent, whichever is longer, prior to dosing
* Known to have received CK-2127107 or tirasemtiv in any previous clinical trial
* Has received or is considering receiving during the course of the study any form of stem cell therapy for the treatment of ALS
* Has received or is considering receiving during the course of the study any form of gene therapy for the treatment of ALS
* Has received or is considering obtaining during the course of the study a diaphragmatic pacing system
* History of substance abuse within the past 2 years
* Use of certain medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD Cytokinetics, Study Director — Cytokinetics
Locations (64):
- United States (47):
  - St. Joseph's Hospital and Medical Center - Barrow Neurological Clinics, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Irvine, Orange, California
  - Forbes Norris MDA/ALS Research Center, San Francisco, California
  - Stanford Hospital and Clinics, Stanford, California
  - University of Colorado Hospital Anschutz Outpatient Pavilion, Aurora, Colorado
  - Hospital for Special Care, New Britain, Connecticut
  - George Washington University Medical Faculty Associates, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Carol & Frank Morsani Center for Advanced Healthcare - University of South Florida, Tampa, Florida
  - Emory Clinic, Atlanta, Georgia
  - Duchossois Center for Advanced Medicine, Chicago, Illinois
  - IU Health Neuroscience Center of Excellence, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University - Outpatient Center, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center/University of Massachusetts Medical School, Worcester, Massachusetts
  - Michigan Medicine, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Saint Louis University, Department of Neurology, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Associates, P.C., Lincoln, Nebraska
  - Hospital For Special Surgery, New York, New York
  - Neurological Institute, Columbia University Medical Center, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Neurosciences Institute, Neurology - Charlotte, Charlotte, North Carolina
  - Duke Neurological Disorders Clinic, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Providence Brain and Spine Institute ALS Center, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center - Clinical Research Center, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - UTHSCSA Medical Arts and Research Center, San Antonio, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - University of Virginia Health System, Charlottesville, Virginia
  - VCU Health - Ambulatory Care Center (ACC), Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - West Virginia University, Dept. of Neurology, Morgantown, West Virginia
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin
- Australia (5):
  - Brain and Mind Centre, The University of Sydney, Camperdown, New South Wales
  - Department of Neurology, Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Perron Institute for Neurological and Translation Science, Nedlands, Western Australia
- Canada (9):
  - University of Calgary, Heritage Medical Research Center, Calgary, Alberta
  - Edmonton Kaye Clinic, Edmonton, Alberta
  - McMaster University Medical Centre, Hamilton, Ontario
  - London Health Sciences Centre University Hospital, London, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Centre de recherche du Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
  - Saskatoon City Hospital, Saskatoon, Saskatchewan
  - CHU de Quebec-Universite Laval, Hopital de l'Enfant Jesus, Québec
- Beaumont Hospital, Dublin, Ireland
- University Medical Center Utrecht, Utrecht, Netherlands
- Hospital San Rafael Servicio de Neurologia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shefner JM, Al-Chalabi A, Andrews JA, Chio A, De Carvalho M, Cockroft BM, Corcia P, Couratier P, Cudkowicz ME, Genge A, Hardiman O, Heiman-Patterson T, Henderson RD, Ingre C, Jackson CE, Johnston W, Lechtzin N, Ludolph A, Maragakis NJ, Miller TM, Mora Pardina JS, Petri S, Simmons Z, Van Den Berg LH, Zinman L, Kupfer S, Malik FI, Meng L, Simkins TJ, Wei J, Wolff AA, Rudnicki SA. COURAGE-ALS: a randomized, double-blind phase 3 study designed to improve participant experience and increase the probability of success. Amyotroph Lateral Scler Frontotemporal Degener. 2023 Aug;24(5-6):523-534. doi: 10.1080/21678421.2023.2216223. Epub 2023 May 30. PMID 37254449
- [Derived] Gebrehiwet P, Meng L, Rudnicki SA, Sarocco P, Wei J, Wolff AA, Chio A, Andrews JA, Genge A, Jackson CE, Lechtzin N, Miller TM, Shefner JM. MiToS and King's staging as clinical outcome measures in ALS: a retrospective analysis of the FORTITUDE-ALS trial. Amyotroph Lateral Scler Frontotemporal Degener. 2023 May;24(3-4):304-310. doi: 10.1080/21678421.2022.2154678. Epub 2022 Dec 12. PMID 36503310
- [Derived] Rudnicki SA, Andrews JA, Genge A, Jackson C, Lechtzin N, Miller TM, Cockroft BM, Malik FI, Meng L, Wei J, Wolff AA, Shefner JM; FORTITUDE-ALS STUDY GROUP. Prescription and acceptance of durable medical equipment in FORTITUDE-ALS, a study of reldesemtiv in ALS: post hoc analyses of a randomized, double-blind, placebo-controlled clinical trial. Amyotroph Lateral Scler Frontotemporal Degener. 2022 May;23(3-4):263-270. doi: 10.1080/21678421.2021.1946083. Epub 2021 Jul 5. PMID 34218726
- [Derived] Shefner JM, Andrews JA, Genge A, Jackson C, Lechtzin N, Miller TM, Cockroft BM, Meng L, Wei J, Wolff AA, Malik FI, Bodkin C, Brooks BR, Caress J, Dionne A, Fee D, Goutman SA, Goyal NA, Hardiman O, Hayat G, Heiman-Patterson T, Heitzman D, Henderson RD, Johnston W, Karam C, Kiernan MC, Kolb SJ, Korngut L, Ladha S, Matte G, Mora JS, Needham M, Oskarsson B, Pattee GL, Pioro EP, Pulley M, Quan D, Rezania K, Schellenberg KL, Schultz D, Shoesmith C, Simmons Z, Statland J, Sultan S, Swenson A, Berg LHVD, Vu T, Vucic S, Weiss M, Whyte-Rayson A, Wymer J, Zinman L, Rudnicki SA. A Phase 2, Double-Blind, Randomized, Dose-Ranging Trial Of Reldesemtiv In Patients With ALS. Amyotroph Lateral Scler Frontotemporal Degener. 2021 May;22(3-4):287-299. doi: 10.1080/21678421.2020.1822410. Epub 2020 Sep 24. PMID 32969758
- [Derived] Shefner JM, Cudkowicz ME, Hardiman O, Cockcroft BM, Lee JH, Malik FI, Meng L, Rudnicki SA, Wolff AA, Andrews JA; VITALITY-ALS Study Group. A phase III trial of tirasemtiv as a potential treatment for amyotrophic lateral sclerosis. Amyotroph Lateral Scler Frontotemporal Degener. 2019;0(0):1-11. doi: 10.1080/21678421.2019.1612922. PMID 31081694

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with familial or sporadic ALS were enrolled at 65 sites in Australia, Canada, Ireland, Netherlands, Spain, and the United States. The first patient was screened on 16 August 2017 and the last patient completed on 07 March 2019.
Pre-assignment Details: Eligible patients were male or female, ≥18 - ≤80 years of age, with familial or sporadic ALS diagnosed for ≤24 months. At screening, patients were to have upright slow vial capacity (SVC) ≥60% of predicted; must have been able to swallow tablets, perform reproducible pulmonary function tests; have normal lab tests; and have a caregiver (if needed).
Groups:
- Placebo: Patients in this group received placebo twice daily for 12 weeks
- Reldesemtiv 150 mg Twice Daily: Patients in this group received 150 mg reldesemtiv twice daily for 12 weeks
- Reldesemtiv 300 mg Twice Daily: Patients in this group received 300 mg reldesemtiv twice daily for 12 weeks
- Reldesemtiv 450 mg Twice Daily: Patients in this group received 450 mg reldesemtiv twice daily for 12 weeks
Period: Overall Study
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 300 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
Started | 115 | 113 (1 patient withdrew consent before study drug dosing and was therefore excluded from safety analysis) | 113 | 117
Completed | 95 | 100 | 97 | 98
Not Completed | 20 | 13 | 16 | 19
Not completed — Adverse Event | 4 | 8 | 7 | 10
Not completed — Death | 1 | 0 | 0 | 1
Not completed — Difficulty Traveling to Clinic Visits | 3 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 1 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Progressive Disease | 4 | 1 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 2 | 0
Not completed — Sponsor Discretion | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 3 | 2 | 1
Not completed — Other | 2 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 300 mg Twice Daily | Reldesemtiv 450 mg Twice Daily | Total
Number analyzed (Participants) | 115 | 112 | 113 | 117 | 457
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.60) | 57.1 (10.91) | 57.8 (10.17) | 60.1 (11.00) | 58.7 (10.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 41 | 42 | 50 | 180
  Male | 68 | 71 | 71 | 67 | 277
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 4 | 2 | 7 | 1 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 1 | 3 | 6 | 0 | 10
  White | 107 | 103 | 100 | 113 | 423
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 3 | 0 | 3 | 9
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 22 | 27 | 27 | 100
  Netherlands | 4 | 2 | 1 | 4 | 11
  United States | 72 | 73 | 71 | 68 | 284
  Ireland | 2 | 2 | 0 | 0 | 4
  Spain | 8 | 9 | 10 | 11 | 38
  Australia | 5 | 4 | 4 | 7 | 20
Time since ALS symptom onset [Mean (Standard Deviation); unit: months] | 22.13 (12.375) | 23.87 (27.503) | 22.52 (14.635) | 22.69 (18.662) | 22.80 (19.080)
Site of symptom onset [Count of Participants; unit: Participants]
  Upper limb | 49 | 52 | 56 | 44 | 201
  Lower limb | 44 | 42 | 40 | 43 | 169
  Bulbar | 22 | 18 | 17 | 30 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Percent Predicted Slow Vital Capacity (SVC)
Description: Slow vital capacity was measured using a spirometer (in units of liters). Following 3 to 5 breaths at rest, patients were instructed to take as deep an inspiration as possible followed by a maximum exhalation (blowing out all the air in their lungs). Values obtained were converted to percent predicted values using the Global Lung Initiative equation (ie, the test result as a percent of predicted values for patients of similar demographic and baseline characteristics [eg, height, age, sex]).
Time Frame: Baseline to Week 12
Population: The outcome measure was analyzed for the Full Analysis Set, which consisted of all randomized patients who received any amount of study drug and had a baseline and at least 1 postbaseline efficacy assessment during double-blind treatment.
Measure: Least Squares Mean (Standard Error); unit: percent predicted
Groups:
- Reldesemtiv 300 mg & 450 mg: For analysis purposes, the results from the reldesemtiv 300 mg group and the 450 mg group were pooled.
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 300 mg Twice Daily | Reldesemtiv 450 mg Twice Daily | Reldesemtiv 300 mg & 450 mg
Number analyzed (Participants) | 114 | 112 | 113 | 117 | 230
percent predicted | -6.46 (0.964) | -4.97 (0.952) | -4.62 (0.963) | -4.58 (0.927) | -4.60 (0.701)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily vs Reldesemtiv 300 mg Twice Daily vs Reldesemtiv 450 mg Twice Daily; The statistical null hypothesis was as follows: there was no assumed dose-response relationship in percent predicted SVC change from baseline to Week 12 among all three active doses and placebo, expressed as: H0: -5 x µ placebo - 1 x µ 150 mg twice daily + 3 x µ 300 mg twice daily + 3 x µ 450 mg twice daily = 0 where µ was the mean of the efficacy endpoint for the designated group; Test type: Superiority; p = 0.1095, Mixed Models Analysis; Analyzed by an MMRM with contrast (-5, -1, 3, 3) to reflect the assumed relationship for the 4 groups: placebo, 150, 300, and 450 mg twice daily; least squares mean treatment difference = 1.61, 95% CI 2-sided [-0.36 to 3.58], Standard Error of Mean 1.003
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.2501, Mixed Models Analysis; Least squares mean difference = 1.49, 95% CI 2-sided [-1.05 to 4.03], Standard Error of Mean 1.291
Statistical Analysis 3: Comparison: Placebo vs Reldesemtiv 300 mg Twice Daily; Test type: Superiority; p = 0.1549, Mixed Models Analysis; Least squares mean difference = 1.84, 95% CI 2-sided [-0.7 to 4.38], Standard Error of Mean 1.29
Statistical Analysis 4: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.1417, Mixed Models Analysis; Least squares mean difference = 1.88, 95% CI 2-sided [-0.63 to 4.38], Standard Error of Mean 1.274
Statistical Analysis 5: Comparison: Placebo vs Reldesemtiv 300 mg & 450 mg; Test type: Superiority; p = 0.0964, Mixed Models Analysis; Least squares mean difference = 1.86, 95% CI 2-sided [-0.33 to 4.05], Standard Error of Mean 1.115

2. Secondary Outcome: Change From Baseline to Week 12 in the ALS Functional Rating Scale - Revised (ALSFRS-R) Total Score
Description: The ALSFRS-R is used to measure the progression and severity of disability in patients with ALS. The ALSFRS-R consists of 12 questions, assessing a patient's capability and independence in functional activities relevant to ALS, categorized in the following 4 domains: gross motor tasks, fine motor tasks, bulbar functions, and respiratory function. Each question is scored from 0 (indicating incapable or dependent) to 4 (normal). The total score ranges from 0 to 48. Higher scores reflect more normal function and lower scores reflect more impaired function.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: change in score
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 300 mg Twice Daily | Reldesemtiv 450 mg Twice Daily | Reldesemtiv 300 mg & 450 mg
Number analyzed (Participants) | 114 | 112 | 113 | 117 | 230
change in score | -3.53 (0.313) | -2.40 (0.311) | -2.62 (0.317) | -2.94 (0.307) | -2.78 (0.228)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily vs Reldesemtiv 300 mg Twice Daily vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.0930, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.56, 95% CI 2-sided [-0.09 to 1.22], Standard Error of Mean 0.335
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.0087, Mixed Models Analysis; Least squares mean difference = 1.13, 95% CI 2-sided [0.29 to 1.97], Standard Error of Mean 0.427
Statistical Analysis 3: Comparison: Placebo vs Reldesemtiv 300 mg Twice Daily; Test type: Superiority; p = 0.0351, Mixed Models Analysis; Least squares mean difference = 0.91, 95% CI 2-sided [0.06 to 1.75], Standard Error of Mean 0.43
Statistical Analysis 4: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.1642, Mixed Models Analysis; Least squares mean difference = 0.59, 95% CI 2-sided [-0.24 to 1.43], Standard Error of Mean 0.425
Statistical Analysis 5: Comparison: Placebo vs Reldesemtiv 300 mg & 450 mg; Test type: Superiority; p = 0.0435, Mixed Models Analysis; Least squares mean difference = 0.75, 95% CI 2-sided [0.02 to 1.48], Standard Error of Mean 0.371

3. Secondary Outcome: Slope of Muscle Strength Mega-score From Baseline to Week 12
Description: A hand-held dynamometer, with a scale of 0 to 300 pounds, was used to measure muscle strength and handgrip strength (bilateral). The muscle groups tested were: elbow flexion, wrist extension, first dorsal interosseous, hip flexion, knee extension, and ankle dorsiflexion; all muscle groups were evaluated bilaterally. For each postbaseline assessment of muscle strength, the percent change from baseline was calculated for each muscle group and handgrip strength, using the following equation: ([postbaseline value - baseline value] / baseline value) × 100. The muscle-strength mega-score was calculated as the average of the changes (ie, percent change from baseline) observed for each of the muscle groups as well as handgrip strength. For this endpoint, negative values indicate a decline in muscle strength.
Time Frame: Baseline to Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: change in mega-score per day
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 300 mg Twice Daily | Reldesemtiv 450 mg Twice Daily | Reldesemtiv 300 mg & 450 mg
Number analyzed (Participants) | 114 | 112 | 113 | 117 | 230
change in mega-score per day | -0.1444 (0.02492) | -0.1198 (0.02463) | -0.1299 (0.02474) | -0.0956 (0.02421) | -0.1127 (0.01731)
Statistical Analysis 1: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily vs Reldesemtiv 300 mg Twice Daily vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.3134, Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Slope difference = 0.0276, 95% CI 2-sided [-0.0261 to 0.0813], Standard Error of Mean 0.02734
Statistical Analysis 2: Comparison: Placebo vs Reldesemtiv 150 mg Twice Daily; Test type: Superiority; p = 0.4824, Mixed Models Analysis; Least squares mean difference = 0.0246, 95% CI 2-sided [-0.0442 to 0.0935]
Statistical Analysis 3: Comparison: Placebo vs Reldesemtiv 300 mg Twice Daily; Test type: Superiority; p = 0.6787, Mixed Models Analysis; Least squares mean difference = 0.0146, 95% CI 2-sided [-0.0544 to 0.0835]
Statistical Analysis 4: Comparison: Placebo vs Reldesemtiv 450 mg Twice Daily; Test type: Superiority; p = 0.1604, Mixed Models Analysis; Least squares mean difference = 0.0488, 95% CI 2-sided [-0.0194 to 0.1171]
Statistical Analysis 5: Comparison: Placebo vs Reldesemtiv 300 mg & 450 mg; Test type: Superiority; p = 0.2966, Mixed Models Analysis; Least squares mean difference = 0.0317, 95% CI 2-sided [-0.0279 to 0.0913]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from administration of the first dose of study drug through 4 weeks after the last dose of study drug.
Description: An AE was treatment-emergent if it started or worsened (eg, increased in severity) during or after the first dose of study drug.
  AEs and SAEs were summarized for the Safety Analysis Set, which consisted of all randomized patients who received at least 1 dose or portion of a dose of study drug.
Arm/Group | Placebo | Reldesemtiv 150 mg Twice Daily | Reldesemtiv 300 mg Twice Daily | Reldesemtiv 450 mg Twice Daily
All-Cause Mortality (participants affected / at risk) | 2/115 | 0/112 | 0/113 | 1/117
Serious Adverse Events (participants affected / at risk) | 10/115 | 8/112 | 8/113 | 8/117
Other Adverse Events (participants affected / at risk) | 95/115 | 99/112 | 97/113 | 107/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=115) | Reldesemtiv 150 mg Twice Daily (N=112) | Reldesemtiv 300 mg Twice Daily (N=113) | Reldesemtiv 450 mg Twice Daily (N=117)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Muscle contractions involuntary (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=115) | Reldesemtiv 150 mg Twice Daily (N=112) | Reldesemtiv 300 mg Twice Daily (N=113) | Reldesemtiv 450 mg Twice Daily (N=117)
Nausea (Gastrointestinal disorders) | 14 (16) | 10 (13) | 13 (14) | 22 (23)
Constipation (Gastrointestinal disorders) | 5 (5) | 7 (8) | 13 (15) | 10 (10)
Diarrhoea (Gastrointestinal disorders) | 8 (8) | 12 (15) | 6 (6) | 4 (4)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2) | 6 (6) | 1 (1)
Headache (Nervous system disorders) | 15 (18) | 16 (18) | 16 (19) | 12 (13)
Dizziness (Nervous system disorders) | 11 (13) | 8 (12) | 11 (13) | 7 (7)
Contusion (Injury, poisoning and procedural complications) | 15 (28) | 8 (15) | 14 (15) | 17 (26)
Post-traumatic pain (Injury, poisoning and procedural complications) | 2 (2) | 6 (8) | 8 (11) | 6 (6)
Skin abrasion (Injury, poisoning and procedural complications) | 5 (7) | 8 (10) | 3 (4) | 5 (7)
Cystatin C increased (Investigations) | 2 (2) | 7 (7) | 9 (9) | 20 (22)
Glomerular filtration rate decreased (Investigations) | 1 (1) | 6 (6) | 6 (6) | 10 (11)
Alanine aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 5 (6) | 11 (14)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (2) | 3 (3) | 9 (11)
Fatigue (General disorders) | 12 (14) | 14 (14) | 19 (20) | 20 (24)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (9) | 4 (5) | 8 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 3 (3) | 6 (7)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (7) | 2 (2) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 9 (9) | 6 (6) | 10 (10) | 9 (9)
Urinary tract infection (Infections and infestations) | 8 (9) | 3 (5) | 5 (5) | 5 (7)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 7 (7) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4) | 3 (3) | 7 (7) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (6) | 6 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (4) | 1 (1) | 2 (3) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/98/NCT03160898/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03160898/SAP_001.pdf